CLINICAL TRIAL: NCT01586806
Title: Postoperative Analgesia Comparing Subsartorial Saphenous Nerve Block With and Without Dexamethasone in ACL Reconstruction
Brief Title: Comparing Subsartorial Saphenous Nerve Blocks With and Without Dexamethasone for Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #2012-002
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-08

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Regional Anesthesia, Saphenous Nerve Block
Keywords: Dexamethasone; Glucocorticoids; Physiological Effects of Drugs; Therapeutic Uses; Anterior Cruciate Ligament Reconstruction; Regional Anesthesia, nerve block; Ultrasonic Imaging; Post-Operative Complications: muscle weakness, pain, nausea and vomiting; Dexamethasone (as local anesthetic additive)
MeSH Terms: conditions — Pain; Nausea; Vomiting | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator)
  Interventions: Drug: Bupivacaine Only
- Dexamethasone 1 mg (Active Comparator)
  Interventions: Drug: Bupivacaine with 1 mg of Dexamethasone
- Dexamethasone 4 mg (Active Comparator)
  Interventions: Drug: Bupivacaine with 4 mg of Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine Only — This is the control treatment arm. Patients will receive an ultrasound-guided saphenous nerve block, consisting of 13 ml of 0.5% bupivacaine (a local anesthetic).
  Arms: Control
Drug: Bupivacaine with 1 mg of Dexamethasone — This is one of two treatment arms. Patients will receive an ultrasound-guided saphenous nerve block, consisting of 13 ml of 0.5% bupivacaine (a local anesthetic), mixed with 1 mg of dexamethasone. Total injection volume will be 15 ml.
  Arms: Dexamethasone 1 mg
Drug: Bupivacaine with 4 mg of Dexamethasone — This is one of two treatment arms. Patients will receive an ultrasound-guided saphenous nerve block, consisting of 13 ml of 0.5% bupivacaine (a local anesthetic), mixed with 4 mg of dexamethasone. Total injection volume will be 15 ml.
  Arms: Dexamethasone 4 mg

SUMMARY:
For patients undergoing Anterior Cruciate Ligament reconstruction surgery, the postoperative period can be a painful experience without adequate pain management. Hence the investigators propose a randomized controlled clinical study, investigating prolonged saphenous nerve blocks. Patients will be randomized to receive saphenous nerve blocks with or without dexamethasone, a corticosteroid used to prolong analgesia.

Depending on the randomized treatment assignment, patients may receive one of the following:

1. 13 ml of 0.5% bupivacaine, a local anesthetic (no dexamethasone);
2. 13 ml of 0.5% bupivacaine mixed with 1 mg of dexamethasone;
3. 13 ml of 0.5% bupivacaine mixed with 4 mg of dexamethasone.

Patients will be followed postoperatively. Following admission to the recovery room, data collectors will ask patients to rate their pain on a scale of 0-10 until discharge. Data collectors will also record patient satisfaction, pain medication use and any side effects experienced (i.e. nausea and vomiting). Patients will then be contacted on postoperative days 1, 2 and 14 and asked questions about their general well-being.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ambulatory surgery for anterior cruciate ligament (ACL) reconstruction with a patella tendon autograft.
* ASA I-III [American Society of Anesthesiologists (ASA) Physical Status classification system]
* BMI < 35
* Smokers included
* Ages 16-65

Exclusion Criteria:

* Patients on steroids or requiring stress dose steroids
* BMI > 35
* Patient refusal
* Allergy to study medications,
* NRS scores > 3 with frequent opioid use (including tramadol) prior to surgery-daily for greater than 3 weeks
* Lower extremity neurological dysfunction
* Diabetic (NIDDM, insulin-dependent and/or oral hypoglycemic dependent)
* Not in included age range (under 16 or over 65 years of age)
* Contraindications to the use of dexamethasone
* Non-English speaking patients. We will be using the Short Form 8 Health Survey, as well as the OR-SDS questionnaire (these are in English; any translations would have to be separately validated).

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2012-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary F. Chisholm, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Vieira PA, Pulai I, Tsao GC, Manikantan P, Keller B, Connelly NR. Dexamethasone with bupivacaine increases duration of analgesia in ultrasound-guided interscalene brachial plexus blockade. Eur J Anaesthesiol. 2010 Mar;27(3):285-8. doi: 10.1097/EJA.0b013e3283350c38. PMID 20009936
- [Background] Cummings KC 3rd, Napierkowski DE, Parra-Sanchez I, Kurz A, Dalton JE, Brems JJ, Sessler DI. Effect of dexamethasone on the duration of interscalene nerve blocks with ropivacaine or bupivacaine. Br J Anaesth. 2011 Sep;107(3):446-53. doi: 10.1093/bja/aer159. Epub 2011 Jun 14. PMID 21676892
- [Background] Portenoy RK, Thaler HT, Kornblith AB, Lepore JM, Friedlander-Klar H, Kiyasu E, Sobel K, Coyle N, Kemeny N, Norton L, et al. The Memorial Symptom Assessment Scale: an instrument for the evaluation of symptom prevalence, characteristics and distress. Eur J Cancer. 1994;30A(9):1326-36. doi: 10.1016/0959-8049(94)90182-1. PMID 7999421
- [Background] Apfelbaum JL, Gan TJ, Zhao S, Hanna DB, Chen C. Reliability and validity of the perioperative opioid-related symptom distress scale. Anesth Analg. 2004 Sep;99(3):699-709. doi: 10.1213/01.ANE.0000133143.60584.38. PMID 15333398
- [Background] Lundblad M, Kapral S, Marhofer P, Lonnqvist PA. Ultrasound-guided infrapatellar nerve block in human volunteers: description of a novel technique. Br J Anaesth. 2006 Nov;97(5):710-4. doi: 10.1093/bja/ael241. Epub 2006 Sep 26. PMID 17005509
- [Background] Akkaya T, Ersan O, Ozkan D, Sahiner Y, Akin M, Gumus H, Ates Y. Saphenous nerve block is an effective regional technique for post-menisectomy pain. Knee Surg Sports Traumatol Arthrosc. 2008 Sep;16(9):855-8. doi: 10.1007/s00167-008-0572-4. Epub 2008 Jun 24. PMID 18574578
- See also: This is the link to Hospital for Special Surgery website. — http://www.hss.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Dexamethasone 1 mg | Dexamethasone 4 mg
Started | 65 | 65 | 65
Completed | 62 | 61 | 63
Not Completed | 3 | 4 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Dexamethasone 1 mg | Dexamethasone 4 mg | Total
Number analyzed (Participants) | 62 | 61 | 63 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (10) | 26 (8) | 27 (10) | 26 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 27 | 19 | 65
  Male | 43 | 34 | 44 | 121
Region of Enrollment [Number; unit: participants]
  United States | 62 | 61 | 63 | 186
Body Mass Index [Mean (Standard Deviation); unit: kg/(m^2)] | 24 (3) | 24 (4) | 25 (3) | 25 (4)

OUTCOME MEASURES:

1. Primary Outcome: Patient-perceived Duration of Analgesia
Description: After discharge, patients will be called and given instructions to help determine length of time of analgesia in the saphenous nerve distribution.
Time Frame: Up to 2 days following surgery
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Control | Dexamethasone 1 mg | Dexamethasone 4 mg
Number analyzed (Participants) | 62 | 61 | 63
hours | 33 [28.4 to 37.3] | 41 [32.4 to 50.9] | 46.5 [35.8 to 48.9]

2. Secondary Outcome: NRS (Numerical Rating Scale) Pain Scores
Description: Patients will be asked to rate, on a scale of 0-10, their pain while at rest. 0 indicates no pain, and 10 indicates the worst pain imaginable.
Time Frame: Postoperative day 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | Dexamethasone 1 mg | Dexamethasone 4 mg
Number analyzed (Participants) | 62 | 61 | 63
units on a scale | 3 [2 to 5] | 3 [1 to 4] | 2 [1 to 4]

3. Secondary Outcome: Patient Satisfaction
Description: Patients will be asked to rate satisfaction on a scale of 0-10 (0=completely dissatisfied, 10=completely satisfied);
Time Frame: Up to 2 days following surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | Dexamethasone 1 mg | Dexamethasone 4 mg
Number analyzed (Participants) | 62 | 61 | 63
units on a scale | 8 [6 to 9] | 8 [6 to 9] | 9 [8 to 10]

4. Secondary Outcome: Postoperative Morphine Consumption
Description: Data collector will record how many opioids (i.e. Percocet, Vicodin) the patient has used since discharge.
Time Frame: Up to 2 days following surgery
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Control | Dexamethasone 1 mg | Dexamethasone 4 mg
Number analyzed (Participants) | 62 | 61 | 63
milligrams | 45 [26.3 to 60] | 30 [22.5 to 60] | 30 [15 to 52.5]

5. Secondary Outcome: Opioid-Related Side Effects (Drowsiness)
Description: Data collector will administer the Opioid-Related Distress Scale (OR-SDS) to determine if patients experience any opioid-related side effects (i.e. drowsiness). The OR-SDS score is on a scale of 0 to 4, with a higher number representing more severe symptoms.
Time Frame: Up to 2 days following surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | Dexamethasone 1 mg | Dexamethasone 4 mg
Number analyzed (Participants) | 62 | 61 | 63
units on a scale | 1.1 [0 to 1.6] | 1 [0 to 1.7] | 0 [0 to 1.4]

ADVERSE EVENTS:
Arm/Group | Control | Dexamethasone 1 mg | Dexamethasone 4 mg
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes